CLINICAL TRIAL: NCT07060261
Title: Prospective Evaluation of Pre-Operative MRI on Margin Status for Transoral Robotic Surgery for HPV+ Tonsillar Squamous Cell Carcinoma
Brief Title: Pre-Op MRI on Margin Status for Transoral Robotic Surgery for HPV+ Tonsillar Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE5325
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-07

CONDITIONS: Human Papilloma Virus Related Carcinoma; Tonsillar Squamous Cell Carcinoma
Keywords: Transoral robotic surgery (TORS); MRI

STUDY DESIGN:
Masking Description: The neuroradiologists will be blinded to each others score
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-operative MRI (Experimental)
  Interventions: Procedure: Transoral robotic surgery+MRI

INTERVENTIONS:
Procedure: Transoral robotic surgery+MRI — During the standard of care MRI, there will be an added T2 and T2 SPACE sequences. These sequences are estimated to take an additional 6 minutes, with no added risk to the patient.

SUMMARY:
This prospective research study aims to see if pre-operative MRI can predict the margin status after transoral robotic surgery (TORS) for human papillomavirus positive (HPV+) tonsillar squamous cell carcinoma (SCC). The pre-operative MRI will have a standard MR neck without and with contrast, with added axial T2 weighted sequence and T2 SPACE sequence through the tonsils. Three neuroradiologists will grade the thickness of the pharyngeal constrictor muscle (the muscle that surrounds the tonsils) on a five-point scale. The study will determine if the pre-operative MRI grading will correlate with positive, insecure (<1mm), or secure (>1mm) margin during TORS surgery for your HPV+ tonsillar SCC.

DETAILED DESCRIPTION:
There has been a marked increase in the incidence on oropharyngeal SCC in recent decades because of the rise of HPV+ disease1-3. Stage I or II tonsillar SCC can be treated by either surgery or radiation with similar good outcomes. For tumors treated surgically, transoral robotic surgery has replaced open surgery due to decreased morbidity and improved local control. It has been shown that margin status of 1.1mm of healthy tissue around the tumor is sufficient for adequate local control. However, approximately 8.1% of the time there is a positive or insecure margin, resulting in added adjuvant radiation and possibly chemotherapy, with increasing morbidity for each added treatment modality.

Therefore, there is a need to determine pre-operatively the chance of positive or insecure margin at surgery to avoid increased morbidity with added adjuvant treatment. Currently, the most commonly used imaging modality is computed tomography (CT) or magnetic resonance imaging (MRI), but this is to rule out absolute contraindications such as internal carotid artery encasement, involvement of the mandibular periosteum, prevertebral fascia/musculature, or masticator space musculature. Recently, a retrospective study used a novel five-point grading scale (1, normal constrictor; 2, bulging constrictor; 3, thinning constrictor; 4, obscured constrictor; and 5, tumor protrusion into the parapharyngeal fat) to evaluate the pharyngeal constrictor muscle, showing that higher scores with obscured constrictor or tumor protrusion into the parapharyngeal fat resulted in increased risk of positive or insecure margin. Given this, there is need for a prospective study to estimate the accuracy of the five-point MRI score with respect to distinguishing patients who go onto have secure surgical margins versus patients who go on to have insecure/positive surgical margins including surgical report of violation of anatomic boundaries (pharyngeal constrictor muscle)

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age.
2. Participants being considered for TORS for HPV+ tonsillar SCC.

Exclusion Criteria:

1. Participants < 18 years of age.
2. Participants who cannot provide informed consent.
3. Participants who do not wish to participate.
4. Vulnerable populations, including but not limited to cognitively impaired persons, pregnant women, and students or house staff under the direct supervision of the investigator.
5. Participants in whom MRI is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy as assessed by 5-point MRI score | Perioperative
  Accuracy will be summarized using the area under the receiver operating characteristics curve (AUC)

SECONDARY OUTCOMES:
Number of Grade 5 cases missed by pre-operative CT versus pre-operative MRI | Perioperative
Percentage of patients who received adjuvant treatment, stratified by MRI grade. | Perioperative
Percentage of participants who received adjuvant therapy, stratified by MRI grade. | Perioperative
Predictive value of tumor size and diffusion/perfusion MRI parameters for post-operative surgical margin status | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided